CLINICAL TRIAL: NCT03600402
Title: Effects and Dose-response of Manual Therapy in the ROM of the Ankle in Older People: Randomized Clinical Trial
Brief Title: Effects and Dose-response of Manual Therapy in the ROM of the Ankle in Older People
Acronym: ANKLE_ROM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, David Hernández, Principal Investigator, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DHG02
Record Dates: First submitted 2018-06-07; First posted 2018-07-26 (Actual); Last update posted 2019-01-04 (Actual); Status verified 2019-01

CONDITIONS: Aging Problems
Keywords: ROM; Manual Therapy; Mobilization; Ankle

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental)
  Interventions: Other: Experimental
- Control Group (Other)
  Interventions: Other: Control

INTERVENTIONS:
Other: Experimental — 6 sessions of ankle manual therapy
  Arms: Experimental Group
Other: Control — 6 sessions of placebo intervention
  Arms: Control Group

SUMMARY:
Limitations of the joint range of the ankle in elderly people is usually common. One of the ways to treat this limitation is through manual therapy, although the effects it produces in dose-response terms are still not well understood. Because of this, this work on the one hand aims to determine the effects and effectiveness of manual therapy and, on the other hand, determine the dose-response necessary for the range of motion of the ankle to improve when applying techniques of manual therapy on the ankle in the older adult.

ELIGIBILITY:
Inclusion Criteria:

* Age
* Ankle dorsiflexion limitation

Exclusion Criteria:

* Do not sign the consent
* No injuries in the foot
* No acute pathology (3 months) in lower limb

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2018-11-12 (Actual); Study Completion 2019-01-03 (Actual)

PRIMARY OUTCOMES:
Active ankle range of movement | Change from baseline to day 1, 3, 5, 8, 10, 12, 19 and 48
  Measurement of the anterior tilt of the tibia during weight bearing with an inclinometer

CONTACTS AND LOCATIONS:
Overall Officials: David Hernández, PT, Principal Investigator — Study Principal Investigator
Locations (1):
- University of Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hernandez-Guillen D, Blasco JM. A Randomized Controlled Trial Assessing the Evolution of the Weight-Bearing Ankle Dorsiflexion Range of Motion Over 6 Sessions of Talus Mobilizations in Older Adults. Phys Ther. 2020 Apr 17;100(4):645-652. doi: 10.1093/ptj/pzaa003. PMID 31944252